CLINICAL TRIAL: NCT06450834
Title: Prospective, Propensity-score Matched Cohort Analysis Evaluating the Use of Ostene Bone Hemostasis Material During Thoracolumbar Decompression, Instrumentation, and Fusion Using a Validated Intraoperative Bleeding Scale
Brief Title: Ostene in Thoracolumbar Decompression and Fusion Evaluated With VIBE
Acronym: Ostene VIBe
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Steven Ludwig, Professor of Orthopaedics, University of Maryland, Baltimore
Other Study IDs: HP-00107929
Record Dates: First submitted 2024-05-28; First posted 2024-06-10 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Intraoperative Complications; Intraoperative Bleeding; Intraoperative Blood Loss; Hemostasis; Blood Transfusion; Postoperative Hemorrhage; Postoperative Complications; Spine Fusion; Thoracolumbar Spine
MeSH Terms: conditions — Intraoperative Complications; Blood Loss, Surgical; Postoperative Hemorrhage; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Ostene: Patients who received Ostene during their thoracolumbar spine surgery
  Interventions: Device: Ostene
- No Ostene: Propensity score matched cohort from previous study that did not receive Ostene during their spine surgery

INTERVENTIONS:
Device: Ostene — Soluble Bone Hemostasis Implant Material
  Groups: Ostene

SUMMARY:
In spine surgery, it is important to try to minimize bleeding. In particular, spine surgery often involves inserting hardware into bone, and/or removing bone in the spine. Because the bone in the spine contains blood vessels, there can often be bleeding from the bone itself that is difficult to stop completely. One way to stop bone bleeding is through the use of wax-like materials, which plug the bleeding bone and act as a physical barrier to stop bleeding. One example is Ostene bone hemostasis material, which has the advantage of being "water soluble", meaning it will dissolve naturally over time. The purpose of this study is to evaluate how well Ostene does at decreasing bleeding, by using a recognized scale called the validated intraoperative bleeding severity scale, abbreviated as "VIBe". In this study, the investigators will record the bleeding severity throughout multiple time points in surgery using this scale, and then the investigators will compare the measurements to patients in the past who did not receive Ostene. Overall, this research will help measure how well Ostene decreases bleeding.

DETAILED DESCRIPTION:
* Patients will be screened prior to surgery for inclusion and exclusion criteria.
* If eligible, patients will be approached in the preoperative area or clinic location to consent or refuse participation in the study.
* Baseline characteristics will be collected via a combination of patient preoperative survey and manual chart review.
* Patients will undergo the normal surgical standard of care, receiving Ostene intraoperatively as determined appropriate by the attending spine surgeon during the procedure.
* It is anticipated that Ostene will be used specifically during the bony work/laminectomy phase preceding decompression. Of note, this material is now considered standard of care by our principal investigator and would be used regardless of study participation.
* Other hemostatic agents will be used according to the typical standard of care.
* A trained research coordinator will be present to determine VIBe scores during 6 key surgical phases: 1) exposure, 2) bony work/laminectomy, 3) decompression, 4) instrumentation, 5) fusion, and 6) closure. Agreement will be obtained from the operating surgeon.
* For all phases, the maximum VIBe score during each phase will be recorded.
* Surgical information will be documented from the operative note.
* Patients will receive the normal standard of care postoperatively including measure(s) of their hemoglobin/hematocrit and postoperative drain output.
* Data on postoperative outcomes/complications will be collected from the electronic medical record.
* A propensity-score matched cohort analysis will be constructed to compare patients who received Ostene to patients who did not receive Ostene (will use data from past study conducted from 2021-April 2023 to construct matched control cohort).

  * There will be no group assignment in this study
  * There will be no placebo group or randomization
  * Patient data from a past study will be used as a control comparator

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 to 88 years old
* Elective thoracolumbar decompression, instrumentation, and fusion procedure
* Open, posterior approach
* Patients included for analysis in a related prior study which had enrollment criteria congruent with the current study

Exclusion Criteria:

* Indication for trauma, tumor, or suspected/confirmed infection
* Emergent triage status
* Anterior or lateral approach
* Minimally invasive approach

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients 18 to 88 years old undergoing elective thoracolumbar decompression, instrumentation, and fusion procedures with an open, posterior approach and without indication for trauma, tumor, or suspected/confirmed infection, emergent triage status, an anterior or lateral approach, or a minimally invasive approach
Sampling Method: Non-Probability Sample
Enrollment: 173 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood transfusion | Intraoperative
  binary and number of units
postoperative blood transfusion | 3 days
  binary and number of units

SECONDARY OUTCOMES:
preoperative hemoglobin/hematocrit | Immediately preoperative
3 days before surgery of preoperative hemoglobin/hematocrit | 3 days
postoperative hemoglobin/hematocrit | 3 days
days after surgery of postoperative hemoglobin/hematocrit | 3 days
postoperative drain output | From the first day postoperatively then measured daily, until the patient is discharged, up to 1 year
  average daily drain output, total drain output
Presence of Deep Vein Thrombosis | From the date of surgery until 1 year follow up appointment
Presence of Pulmonary Embolism | From the date of surgery until 1 year follow up appointment
Presence of postoperative complication requiring medical intervention | From the date of surgery until 1 year follow up appointment
length of stay | From the date of surgery until discharge up to 1 year
30-day readmissions | readmission within 30 days
30-day reoperations | reoperation within 30 days
30-day emergency department visits | ED visits within 30 days
cost | From the date of surgery until discharge up to 1 year
  total hospital billing for procedure and total episode of stay and/or insurance reimbursement amount

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share IPD data with any other researchers.